CLINICAL TRIAL: NCT04137406
Title: Role of SIRT1 in Regulation of Epithelial-to-mesenchymal Transition in Breast Cancer Lymph Nodes Metastasis for Luminal A Subtype
Brief Title: Role of SIRT1 in Regulation of Epithelial-to-mesenchymal Transition in Breast Cancer Lymph Nodes Metastasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Luminal A sirt1
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer; Lymph Node Metastases
Keywords: Luminal A breast cancer; Sirt 1; lymph node metastasis; EMT
MeSH Terms: conditions — Breast Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Paraffin section, immunohistochemical staining
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- T1 tumor with lymph node metastasis: patients with T1 tumor and lymphnode positive
- T2 or T3 tumor with lymph node negative: patients with T2 or T3,lymph node negative

SUMMARY:
Luminal A breast cancer is a kind of breast cancer with low rate lymph node metastasis and good survival. But in clinical practice, Luminal A breast cancer can present with early, unexpected lymph node metastasis some time, indicates poor survival. Silent information regulator 2 homolog 1 (SIRT1) plays a different role in breast cancer with different molecular typing. Previous study supports a role of SIRT1 protein as tumor suppressor in Luminal A breast cancer, in association with apoptosis-related proteins. The epithelial-to-mesenchymal transition(EMT) process results in loss of cell-cell adhesion, increased cell mobility, and is crucial for enabling the metastasis of cancer cells. But no similar study in Luminal A breast cancer. Hence, this study will 1) investigate the expression pattern of SIRT1 in primary tumor and lymph node metastasis; 2) investigate the different expression pattern of SIRT1 in T2/T3 , lymph node negative tumor and T1, lymph node positive tumor; 3) investigate potential role of SIRT1 enzyme in regulating cell migration and invasion in Luminal A breast cancer cells.

DETAILED DESCRIPTION:
The study has three parts.

1. In large specimens of human Luminal A breast cancer with T1 tumor and positive axillary lymph node, study the difference expression of SIRT1 and related p53, Bcl-2, autophagy-related protein caspase-3, apaf-1 between primary tumor and lymph node metastases. Collect 50 pairs of T1 primary tumors and corresponding metastatic lymph node specimens. Using immunohistochemistry, anti-SIRT1, p53, Bcl-2, caspase-3 and apaf-1 antibody staining to identify the expression of above proteins in the primary tumor and lymph node metastases.
2. Eighty patients with Luminal type A breast cancer (T1N+) were enrolled in this study. At the same time,eighty patients were enrolled in the paraffin-embedded specimens of the patients with T2N+ and T3N+,too. And all patients were followed up. Immunohistochemical staining with anti-SIRT1, p53, Bcl-2, caspase-3, apaf-1, E-cadherin, N-cadherin, Vimentin antibodies to determine the relationship between above protein expression and routine clinicopathological and survival.
3. Explore the involvement of SIRT1 in hormone receptor-positive human breast cancer cells at the cellular level. The molecular mechanism of EMT-related protein regulation, which affects the proliferation, invasion and metastasis of tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* Invasive breast cancer Luminal A subtype T1 and lymph node positive or T2/T3 with negative lymph node

Exclusion Criteria:

* Missing clinical pathology data

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all the patients have invasive breast cancer with luminal A subtype group 1: T1 and lymph node positve group 2: T2/T3 with negative lymph node
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Protein expression difference | 2020-2
  the different of sirt1 expression between T1N+ tumor and T2N0/T3M0 tumor

SECONDARY OUTCOMES:
survival | 2021-2
  the relationship of sirt1 expression level and survival

CONTACTS AND LOCATIONS:
Overall Officials: shu wang, Doctor, Study Director — Peking University People's Hospital
Locations (1):
- Peking university people's hospital, Beijing, Beijing Municipality, China